CLINICAL TRIAL: NCT02768636
Title: Can Omega-3 Improve Heart Rate Variability Measurement?
Acronym: HRV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vachira Phuket Hospital (Other)
Responsible Party: Principal Investigator, Jessada Chungpaibulpatana, Tappana Sumpatanarax, Director, Principal investigator; Co-investigator, Vachira Phuket Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VPH2016001
Record Dates: First submitted 2016-05-03; First posted 2016-05-11 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Individuality
Keywords: Omega-3, ANS, HRV, SDNN
MeSH Terms: interventions — Docosahexaenoic Acids; Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Before and after omega-3 used (Experimental): Before and after omega-3 used
  Interventions: Dietary Supplement: Omega-3

INTERVENTIONS:
Dietary Supplement: Omega-3 — Omega-3 or Fish oil (1000 mg.) is taken for one capsule a day in 30 days duration. Heart rate variability is tested before at starting day and later follow up it again in the next 30 days appointment.
  Other Names: Fish oil

SUMMARY:
Heart rate variability can represent physiological and psychological levels via sympathetic and parasympathetic variables on autonomic nervous function. Omega-3 has shown that it can effect on physiological and psychological with many good results. The pathways to explain about its effect had been studied in many contexts. Effect to autonomic nervous function by Omega-3 is our interesting question.

DETAILED DESCRIPTION:
Heart Rate Variability (HRV). HRV has two domains, time domain and frequency domain. SDNN (Standard Deviation Normal to Normal) is the first time domain. In healthy state, the signal is more diversity and SDNN is high. Decrease of SDNN means that ability to maintain homeostasis is reduced. It is shown while a person is in any disease state. Significant decreasing of HRV is an indicator for general health. PSI (Physical Stress Index) is the pressure loaded state due to overloaded physical activity and heart rate is increasing. Total power (TP), Very low frequency (VLF), Low frequency (LF), High frequency (HF), normalized Low frequency (nLF, LF norm) = LF/(LF +HF), normalized High frequency (nHF, HF norm) = HF/(LF+HF) and Low frequency to High frequency ratio (LF/HF) are frequency domain. Mean Heart rate (MHR) is also an indicator representing autonomic function.

Range of study: It will be done during April - May 2016.

Population Enrollment and recruitment was done by selected volunteers for our 100 participants.

Investigator: Training investigators were selected from psychologists, technicians, nurses, medical students and hospital health colleagues. Certified attending the class of training, assessment and evaluation was done before study.

Maneuver: Instruments were questionnaires and HRV measurements by SA-3000P. Fast Fourier Transformation method (FFT) was applied underlying it. Finger probe was used by five minutes with comfort sitting upright position. Normal respiration and not heavy pay attention in the monitor by looking to the wall. Enough sleeping in the night before study and no take coffee, drugs, alcohol or smoking two hours before study.

Variables: HRT, Heart rate; SDNN, Standard deviation of normal to normal interval; RMSSD, the square root of the mean squared differences of successive NN intervals; PSI, Physical stress index; ApEn, Approximate Entropy; SRD, Successive R-R interval difference; TSRD, Total SRD;TP, Total power; VLF, Very low frequency; LF, Low frequency; HF, High frequency; nLF, normalized LF; nHF, normalized HF.

Statistical analysis: We use descriptive study and report it in percents, means, standard deviations, medians, inter quartiles ranges. Independent t-test and ANOVA were used in parametric test. Pearson Chi-square Test, Mann-Whitney U Test, Kruskal-Wallis Test, Kolmogorov-Smirnov Z Test, Wald-Wolfowitz Test were used in nonparametric test. Significance of statistical analysis was 0.05 or 95% confidence interval. Units of SDNN is millisecond (ms) and TP, VLF, LF, HF are square of millisecond (ms2) multiply by 100. Comparative study (before and after) will use paired t-test or non-parametric (McNemar test, Sign test or Wilcoxon).

Conflict of interest: We receive these products (Omega-3, Fish oil) from Starlab company and this manufacturing will be stop to produce this agent in this April because of high business competition. They donate the remaining products for this research.

ELIGIBILITY:
Inclusion Criteria:

1. Aged group is 18-65 years old
2. Understanding communication
3. Normal electrocardiogram
4. Allowance by their physicians
5. No disturbance with their regular treatments

Exclusion Criteria:

1. Abnormal bleeding tendency problems
2. Non-understanding communication
3. No enough time persons
4. No information allowance
5. Complicated illnesses conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate Variability assessed using the SA-3000P | Baseline and 30 days
  Comparative participants' Heart rate variability study will be done before and after 30 days treated with Omega-3. Instruments were questionnaires and HRV measurements by SA-3000P. Fast Fourier Transformation method (FFT) was applied underlying it. Finger probe was used by five minutes with comfort sitting upright position. Variables: HRT (BPM), Heart rate; SDNN (ms), Standard deviation of normal to normal interval; RMSSD (ms), the square root of the mean squared differences of successive NN intervals; PSI (No scale), Physical stress index; ApEn (No scale), Approximate Entropy; SRD (No scale), Successive R-R interval difference; TSRD (No scale), Total SRD; TP (ms^2), Total power; VLF (ms^2), Very low frequency; LF (ms^2), Low frequency; HF (ms^2), High frequency; nLF (n.u.), normalized LF; nHF (n.u.), normalized HF, LF/HF, Low frequency/ High frequency

CONTACTS AND LOCATIONS:
Overall Officials: Jessada Chungpaibulpatana, MD., Study Director — Director
Locations (2):
- Thailand (2):
  - Vachira Phuket Hospital, Phuket, Phuket
  - Vachira Phuket, Phuket, Phuket

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Asterios P. Deligiannis. The Effects of Exercise Training on Cardiac Autonomic Nervous Activity. Available from — http://www.fac.org.ar/tcvc/llave/c243/deligian.PDF
- See also: Front Physiol. 2011; 2: 84. published online 2011 Nov 16. Prepublished online 2011 Oct 4.doi: 10.3389/fphys.2011.00084 Available from — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3217222/
- See also: Cicka, Danielle, "The Effect of Omega-3 Fatty Acids on Heart Rate Variability, Coronary Heart Disease, and Depression" (2013). Washington University Undergraduate Research Digest, Volume 9, Issue 1. Available from — http://openscholarship.wustl.edu/vol9_iss1/25
- See also: K. Connor, W. Zhang, V. Payne, V. Payne, L. Watkins, D. Watkins. Neuropsychopharmacology; 2005. Available from — http://www.nordicnaturals.com/images/researchImages/Connor_DukeABSTRACT.pdf
- See also: Dariush Mozaffarian, Phyllis K. Stein, Ronald J. Prineas, David S. Siscovick. Circulation. 2008;117:1130-1137. Available from — http://circ.ahajournals.org